CLINICAL TRIAL: NCT00889980
Title: Sentinel Node and Non-Sentinel Lymph Nodes (SLN and Non-SLN) Procurement From Melanoma Subjects for Molecular Profiling Analysis
Brief Title: Melanoma Molecular Profiling Analysis
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, John Kirkwood, MD, University of Pittsburgh
Other Study IDs: 07-133
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Lymph nodes (less than 20% of any node), blood will be drawn at the pre study visit (serum and peripheral blood mononuclear cells) and appropriate lineage control tissue will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Melanoma: Patients with primary melanoma
  Interventions: Other: Biospecimen banking

INTERVENTIONS:
Other: Biospecimen banking — SLN and one non-SLN (8mm and larger in longest dimension). fourteen 10cc tubes or a total of 140mL of blood will be collected from subjects weighing over 102.6 pounds. If the subject weighs less than 102.6 pounds, the amount of blood drawn will be based on exact body weight. The amount of blood drawn will be no more than 3mL/kg of body weight.

SUMMARY:
There is a significant need to develop new and more effective ways to treat melanoma that will decrease patient morbidity and mortality. This protocol intends to collect and process a portion (< 20% of any node) of lymph nodes from melanoma patients undergoing routine surgical SLN resection: the SLN(s) and 1 adjacent non-SLN(s) are planned for study. In addition, blood will be drawn at the pre study visit (serum and peripheral blood mononuclear cells) and appropriate lineage control tissue will be collected. Material only from already-indicated and planned procedures as part of standard medical care will be used. The main goal of this study will be to properly collect and process material to be analyzed and explore the molecular features melanoma biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Primary melanoma with the following Breslow thickness and stage

  * ≥ 2 mm with ulceration, T3b
  * ≥ 4 mm without (T4a) or with (T4b) ulceration
  * Patients with a biopsied tumor that has not been widely resected will also be eligible for study according to the above-specified criteria for tumor thickness and stage.
* Age 12 years or older.
* Patients must have documented hemoglobin level of 10g/dL or higher. This can be drawn on the day of consent, or be documented from a previous visit within the past 30 days
* Subjects must have provided written, informed consent prior to any study procedures: collection of blood and LN tissue specimens for this protocol.

Exclusion Criteria:

* Serious illnesses that may be considered a contraindication to surgery as determined by the physician investigator. If a subject is cleared for surgery as clinically indicated (wide excision of the primary melanoma and sentinel lymph node biopsy), subject would be eligible.
* Any significant psychiatric disease, medical intervention, or other condition, which in the opinion of the Principal Investigator or Co-Investigators, could prevent adequate informed consent or compromise participation in the clinical trial.
* Active infection or antibiotics within one-week prior to study
* Systemic steroid or other immunosuppressive therapy administered for more than 10 days within 4 weeks of enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Melanoma patients
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2008-05; Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Molecularly characterize the regional nodal status of positive and negative SLNs (SLN+ and SLN-) in patients undergoing SLN mapping and dissection for routine staging of melanoma. | 2 years

SECONDARY OUTCOMES:
Biomarkers differentially expressed between SLN+ and SLN- specimens, molecular profiling the SLN+ node and adjacent non-SLN, and if association exists between specific gene signatures for positive and negative SLN and clinical outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States